CLINICAL TRIAL: NCT00805870
Title: The Effects of High Dose Fish Oil Supplementation on Delayed Onset Muscle Soreness and Inflammatory Markers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Christopher Cheatham, Chair and Associate Professor, Western Michigan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-02-31
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Muscle Damage; Muscle Inflammation
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Omacor; wheat germ oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish Oil (Experimental): Lovaza, 3 grams/day for 65 days
  Interventions: Drug: Lovaza (omega-3-acid ethyl esters)
- Control (Placebo Comparator): Wheat Germ Oil, 3 grams/day for 65 days
  Interventions: Drug: Wheat Germ Oil

INTERVENTIONS:
Drug: Lovaza (omega-3-acid ethyl esters) — Lovaza, 3 grams per day for 65 days
  Arms: Fish Oil
Drug: Wheat Germ Oil — Wheat germ oil, 3 grams/day for 65 days
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of fish oil supplementation (Lovaza, GlaxoSmithKline) on muscle strength, muscle soreness and inflammation following exercise.

DETAILED DESCRIPTION:
When a person exercises at a high intensity or starts a new exercise program, muscle soreness will develop. Muscle soreness that peaks between 24-72 hours after exercise and diminishes in 5-7 days is characterized as delayed onset muscle soreness (DOMS). DOMS is associated with the eccentric phase of exercise, where the muscle is actively creating force while lengthening. The onset of muscle soreness is part of an inflammatory response due to the muscular damage caused by the exercise.

Research has shown that fish oils have anti-inflammatory properties. Direct intake of various polyunsaturated fatty acids (PUFA) alters the cell membrane fatty acid composition, which, in turn modulates cell/tissue response to infection, injury and inflammatory events. These properties may be beneficial to relieve muscle soreness.

Therefore, the purpose of this study is to determine the effects of fish oil supplementation (Lovaza, GlaxoSmithKline, 3 grams per day for 65 days) on muscle strength, muscle soreness and inflammation following exercise.

Participants will be randomly assigned to one of two groups: Lovaza (3 grams/day) or placebo. Participants will consume either the Lovaza or the placebo for 65 consecutive days. On Day 60, participants will have baseline measurements of muscle strength, muscle soreness, creatine kinase activity, and muscle inflammatory marker assessed. Participants will then perform eccentric exercise on an isokinetic dynamometer using the quadriceps muscles in order to induce muscle soreness. On each of Days 61-65, muscle strength, muscle soreness, creatine kinase activity, and muscle inflammatory markers will again be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, free of disease
* Must be able to swallow capsules
* Free of orthopedic or muscular injuries
* Recreationally active
* Prior consumption of fish and corn with no adverse reactions

Exclusion Criteria:

* Use of non-steroidal anti-inflammatory drugs (NSAIDS) or topical analgesics during study enrollment
* Pregnant or nursing
* Food allergy to fish or any components of the pills which includes alpha tocopherol, partially hydrogenated vegetable oils including soybean oils and gelatin and glycerol or wheat germ oil
* Competitive athlete or physically active more than 10 hours per week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Cheatham, Ph.D., Principal Investigator — Western Michigan University
Locations (1):
- Western Michigan University, Kalamazoo, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fish Oil | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.9 (1.7) | 23.4 (2.3) | 22.7 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength
Description: Quadriceps muscle strength is the maximal amount of force that the quadriceps muscles can produce during isometric knee extension exercise.
Time Frame: 6 days
Population: Number of subjects that completed the protocol. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Fish Oil: 3 grams/day of fish oil for 65 days
- Control: 3.45 grams/day of wheat germ oil for 65 days
Arm/Group | Fish Oil | Control
Number analyzed (Participants) | 10 | 10
lbs | 151 (6) | 160 (8)
Statistical Analysis 1: Comparison: Fish Oil vs Control; Null hypothesis is that no difference is observed in quadriceps muscle strength between the fish oil and control groups; Test type: Superiority or Other; p > 0.05, ANOVA; Mean Difference (Net) = 8.271, 95% CI 2-sided [-63.521 to 46.978], Standard Error of Mean 26.298

2. Primary Outcome: Muscle Soreness of the Quadriceps Using an Algometer Strain Gauge
Description: The required amount of force applied to the quadriceps to elicit pain or discomfort.
Time Frame: 6 days
Population: Number of subjects that completed the protocol. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Fish Oil | Control
Number analyzed (Participants) | 10 | 10
lbs | 14.62 (0.47) | 16.46 (0.37)
Statistical Analysis 1: Comparison: Fish Oil vs Control; Null hypothesis is that there is no difference in the amount of force applied to the quadriceps to elicit pain or discomfort between the fish oil and control groups; Test type: Superiority or Other; p > 0.05, ANOVA; Mean Difference (Net) = -1.845, 95% CI 2-sided [-4.823 to 1.132], Standard Error of Mean 1.417

3. Primary Outcome: Creatine Kinase Activity Measured in Blood
Description: Creatine kinase activity is an indirect indicator of muscle damage.
Time Frame: 6 days
Population: Number of subjects that completed the protocol. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fish Oil | Control
Number analyzed (Participants) | 10 | 10
IU/L | 110.20 (11.81) | 167.21 (15.18)
Statistical Analysis 1: Comparison: Fish Oil vs Control; Null hypothesis is that there is no difference in creatine kinase activity between the fish oil and the control groups; Test type: Superiority or Other; p > 0.05, ANOVA; Mean Difference (Net) = -57.015, 95% CI 2-sided [-156.373 to 42.344], Standard Error of Mean 47.093

4. Primary Outcome: Interleukin-6 Measured in Blood
Description: Interleukin-6 is an indirect indicator of muscle inflammation.
Time Frame: 6 days
Population: Number of subjects that completed the protocol. Analysis was per protocol
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fish Oil | Control
Number analyzed (Participants) | 10 | 10
pg/mL | 0.23 (0.07) | 0.21 (0.05)
Statistical Analysis 1: Comparison: Fish Oil vs Control; The null hypothesis is that there is no difference in interleukin-6 concentration between the fish oil and control groups; Test type: Superiority or Other; p > 0.05, ANOVA; Mean Difference (Net) = 0.022, 95% CI 2-sided [-0.374 to 0.417], Standard Error of Mean 0.188

ADVERSE EVENTS:
Arm/Group | Fish Oil | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes